CLINICAL TRIAL: NCT01625936
Title: Phase 1b Study Of CRLX 101 (Cerulean) In Combination With Bevacizumab In The Treatment Of Patients With Advanced Renal Cell Carcinoma
Brief Title: CRLX101 Plus Bevacizumab in Advanced RCC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: UPCC 02812
Record Dates: First submitted 2012-06-20; First posted 2012-06-22 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Renal Cell Carcinoma
Keywords: metastatic; locally advanced; unresectable
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasm Metastasis | interventions — IT-101; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: CRLX101 (Cerulean) — CRLX101 is an innovative tumor-targeting nanopharmaceutical.
Drug: Bevacizumab

SUMMARY:
This is a Phase 1b, dose escalation study of the investigational agent, CRLX101, given in combination with Bevacizumab in patients with advanced renal cell carcinoma. The purpose of this study is to determine the initial safety and effectiveness of this agent in combination with Bevacizumab. The investigators are also trying to determine the best dose level of CRLX101 to give in combination with bevacizumab. About 22 subjects will be enrolled in this study at the University of Pennsylvania.

DETAILED DESCRIPTION:
This is a Phase 1b, dose-escalation study of the investigational agent, CRLX101, given in combination with Bevacizumab in patients with advanced renal cell carcinoma. The purpose of this study is to determine the initial safety and effectiveness of this agent in combination with Bevacizumab. The investigators are also trying to determine the best dose level of CRLX101 to give in combination with Bevacizumab. About 22 subjects will be enrolled in this study at the University of Pennsylvania. This study also involved two sub-studies that will be conducted in a select set of study subjects. This includes investigational cG250 PET/CT scans and paired bone marrow biopsy/aspirate assessments. The IND being requested from the FDA for this study will cover both the use of CRLX 101 as well as the use cG250 in the study sub-study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed metastatic or locally advanced renal cell carcinoma that is unresectable.
* Patients must have disease that is evaluable by the Response Evaluation Criteria in Solid Tumors guidelines (RECIST), v1.1. Disease sites must be assessed within 4 weeks of study entry.
* Patients must have been treated with at least one prior conventional molecularly targeted therapy in a non-adjuvant setting. Conventional molecularly targeted therapy will be defined as including pazopanib, sorafenib, sunitinib, temsirolimus, axitinib, or everolimus.
* A two week wash out is required between the last dose of molecularly targeted therapy and baseline correlative studies (124I-cG250 PET/CT and bone marrow biopsy). If no baseline correlative studies will be performed, a wash out of 1 week will be required prior to the commencement of study therapy. Toxicities from prior therapy must be resolved to grade 1 or less prior to the start of study therapy.
* Patients may have been treated with surgery or not (i.e., cytoreductive nephrectomy not required), radiation therapy, chemotherapy, cytokine therapy including interferon alpha and interleukin-2.
* Patients with treated brain or spinal-associated metastases are eligible but must have concluded dexamethasone therapy and be considered neurologically stable.
* Age greater or equal to 18 years.
* ECOG performance status less than 1 (Karnofsky greater than 70%)
* Life expectancy greater than 3 months.
* Patients must have normal organ and marrow function
* The effects of CRLX101 and bevacizumab on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal, barrier method, abstinence) prior to study entry, for the duration of study participation, and 4 months after completion of administration of this combination therapy. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform the treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and for 4 months after completion of administration of this combination therapy.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had conventional chemotherapy or radiotherapy within 2 weeks prior to entering the study or those who have not yet recovered to grade 1 or less prior treatment-related adverse events.
* Patients who have had major surgery within the last 4 weeks.
* Prior treatment with bevacizumab or topoisomerase I therapy.
* Patients who are receiving any other investigational therapeutic agent.
* History of allergic reactions attributed to any of the experimental compounds examined in this study.
* No other active malignancy (inactive / without progression for at least 6 months and no progression anticipated).
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active serious infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* History of non-healing wounds or ulcers.
* Pregnant or nursing patients as stated above. Agents examined in this clinical trial carry the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with study agents, breastfeeding should be discontinued if the mother is treated on study.
* Bevacizumab has been associated with the development of treatment-related hypertension that can become urgent or emergent. Evidence of uncontrolled hypertension in patients prior to study enrollment will preclude enrollment onto this study until blood pressure is controlled. Uncontrolled hypertension is defined as the presence of systolic blood pressure greater or equal to 150 mmHg or diastolic blood pressure greater or equal to 100 mmHg measured on two separate occasions.
* Patients with known HIV or with solid organ transplant (because of potential additional risk for cytopenias).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2012-06; Primary Completion 2017-07-01 (Actual); Study Completion 2018-07-16 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Naomi M Haas, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States